CLINICAL TRIAL: NCT01615718
Title: Effects of Non-invasive Neurostimulation Methods on Motor Function in Parkinson's Disease Patients.
Brief Title: Non-invasive Neurostimulation in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Highland Instruments, Inc. (Industry)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-p-001120; 1R44NS080632-01 (NIH)
Record Dates: First submitted 2012-05-30; First posted 2012-06-11 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Parkinson's Disease
Keywords: noninvasive stimulation; motor function; transcranial stimulation; transcranial ultrasound; brain stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- Active Electrical Stim/Active Ultrasound (Experimental): Subjects will undergo active low-intensity transcranial electrical stimulation in conjunction with active transcranial ultrasound for 20 minutes.
  Interventions: Procedure: low-intensity transcranial electrical stimulation; Procedure: transcranial ultrasound
- Sham Electrical Stim/Sham Ultrasound (Sham Comparator): Subjects will undergo sham (placebo) low-intensity transcranial electrical stimulation in conjunction with sham transcranial ultrasound for 20 minutes.
  Interventions: Procedure: low-intensity transcranial electrical stimulation; Procedure: transcranial ultrasound
- Active Electrical Stim/Sham Ultrasound (Active Comparator): Subjects will undergo active low-intensity transcranial electrical stimulation in conjunction with sham (placebo) transcranial ultrasound for 20 minutes.
  Interventions: Procedure: low-intensity transcranial electrical stimulation; Procedure: transcranial ultrasound
- Sham Electrical Stim/Active Ultrasound (Active Comparator): Subjects will undergo sham (placebo) low-intensity transcranial electrical stimulation in conjunction with active transcranial ultrasound for 20 minutes.
  Interventions: Procedure: low-intensity transcranial electrical stimulation; Procedure: transcranial ultrasound

INTERVENTIONS:
Procedure: low-intensity transcranial electrical stimulation — Subjects will undergo 20 minutes of low-intensity transcranial electrical stimulation of up to 2mA. During active stimulation, the current will be active for 20 minutes - however, during sham stimulation (placebo) the current will not be active for the full 20 minutes.
Procedure: transcranial ultrasound — Subjects will undergo 20 minutes of transcranial ultrasound. During active stimulation, the ultrasound will be active for 20 minutes - however, during sham stimulation (placebo) the ultrasound will not be active for the full 20 minutes.

SUMMARY:
In this study, the investigators aim to investigate the effects of non-invasive neurostimulation - low-intensity transcranial electrical stimulation in conjunction with transcranial ultrasound (TUS)- on the motor symptoms associated with Parkinson's disease. The investigators want to see if there is a difference between active and sham stimulation on these motor symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of PD diagnosis from their clinician by either a letter or verification through their medical record
* Research criteria of "possible" or "probable" PD, as defined by Gelb et al (Gelb D, Oliver E, Gilman S. Diagnostic Criteria for Parkinson Disease. Arch Neurol.1999;56:33-39)[1]
* Age 40 or over;
* Taking stable medications for at least 30 days

Exclusion Criteria:

* Features suggestive of other causes of parkinsonism/Parkinson's-plus syndromes;
* History of deep brain stimulation or ablation surgery, mass brain lesions;
* History of schizophrenia, schizoaffective disorder, other psychosis, episode of bipolar illness, alcohol/drug abuse within the past year;
* Need for rapid clinical response due to conditions such as initiation, psychosis, or suicidal;
* Contraindications to transcranial brain stimulation or TUS, i.e. metal in the head, implanted brain medical devices, etc;
* Unstable medical conditions (e.g. uncontrolled diabetes, uncompensated cardiac issues, heart failure, pulmonary issues, or chronic obstructive pulmonary disease);
* Pregnancy.
* Epilepsy or disorders that increase likelihood of seizures including: moderate or severe traumatic brain injury, congenital birth defects leading to seizures, brain tumor, metabolism disorders associated with seizures, and nonlacunar stroke.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-09; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Changes in Motor Function | Measured for approximately 2 months
  We will measure motor symptoms using the Unified Parkinson's Disease Rating Scale (UPDRS), bradykinesia tests and walking tests. We will assess the changes in these scales from baseline.

SECONDARY OUTCOMES:
Safety | Measured for approximately 2 months
  We will measure safety using a battery of electrophysiology, cognitive and neurological safety markers. We will use the Scales for Outcomes in PD-Cognitive (SCOPA-COg), the n-back working memory test, adverse effects questionnaire, electroencephalography (EEG) and a standardized neurological exam
Neurophysiological Changes | Measured for approximately 2 months
  We will also use transcranial magnetic stimulation (TMS) and Doppler Ultrasound to assess electrophysiology and cerebral bloodflow markers.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wagner, PhD, Principal Investigator — Highland Instruments, Inc.; Felipe Fregni, MD, PhD, MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States